CLINICAL TRIAL: NCT04759144
Title: A Randomised Crossover Study Comparing Hybrid Closed-loop Insulin Delivery Using Ultra-rapid Acting Insulin to Hybrid Closed-loop Insulin Delivery Using Standard Rapid-acting Insulin in Children With Type 1 Diabetes in the Home Setting (FAST-Kids)
Brief Title: FASter Insulin in Closed-loop Technology in Children
Acronym: FAST-Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Study Director, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FAST-Kids
Record Dates: First submitted 2021-02-13; First posted 2021-02-18 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Faster insulin aspart; Closed loop insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Device: CamAPS FX
  The automated closed loop system (CamAPS FX) will consist of:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data.
  Treatment: Two insulins will be used
  * Faster insulin aspart (Fiasp)
  * Standard insulin aspart (Novorapid)
Who Masked: Participant, Care Provider, Investigator
Masking Description: An unmasked member of staff will undertake randomisation. The participants and the clinical staff will be blind to allocated treatment sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faster insulin aspart with hybrid closed-loop insulin delivery (Active Comparator): Unsupervised home use of hybrid closed-loop insulin delivery with faster insulin aspart for 8 weeks.
  Intervention: Use of faster insulin aspart with hybrid closed-loop insulin delivery
  Interventions: Device: CamAPS FX using faster insulin aspart
- Standard insulin aspart with hybrid closed-loop insulin delivery (Active Comparator): Unsupervised home use of hybrid closed-loop insulin delivery with standard insulin aspart for 8 weeks.
  Intervention: Use of standard insulin aspart with hybrid closed-loop insulin delivery
  Interventions: Device: CamAPS FX using standard insulin aspart

INTERVENTIONS:
Device: CamAPS FX using faster insulin aspart — CamAPS FX closed loop system comprises:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data
  Arms: Faster insulin aspart with hybrid closed-loop insulin delivery
Device: CamAPS FX using standard insulin aspart — CamAPS FX closed loop system comprises:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data
  Arms: Standard insulin aspart with hybrid closed-loop insulin delivery

SUMMARY:
The main objective of this study is to determine whether 24/7 hybrid closed-loop insulin delivery under free living conditions applying faster insulin aspart (FiAsp) is superior to 24/7 hybrid closed-loop insulin delivery applying standard insulin aspart in very young children with type 1 diabetes.

The closed-loop system consists of three components: the continuous glucose monitor (CGM), the insulin pump and a smartphone Application, or App, that translates, in real-time, sensor glucose levels received from the glucose monitoring device and calculates the amount of insulin to be delivered by the coupled insulin pump.

This is a double-blind, multi-centre, randomised, crossover design study, involving a run-in period followed by two 8-week study periods during which glucose levels will be controlled by a hybrid closed-loop system using either standard insulin aspart or faster insulin aspart in random order.

Participants aged 2-6 years with type 1 diabetes on insulin pump therapy will be recruited through paediatric diabetes outpatient clinics at participating clinical centres. Enrolment will target up to 30 children (aiming for 6-14 participants per centre) to allow for dropouts during run-in.

Prior to the use of study devices, participants and parents/guardians will receive appropriate training by the research team on the safe use of the study pump and CGM device, and the hybrid closed-loop insulin delivery system. Parents/guardians at nursey/school may also receive training by the study team if required. Participants will have regular contact with the study team during the study including 24/7 telephone support. Parents/guardians will be asked to complete validated questionnaires at the start and end of the study to assess quality of life measures including sleep.

The primary outcome is the between group difference in time spent in target range between 3.9 and 10.0 mmol/l as recorded by CGM during the study. Secondary outcomes are time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics. Safety evaluation comprises assessment of the frequency and severity of hypoglycaemic episodes and diabetic ketoacidosis (DKA).

DETAILED DESCRIPTION:
Purpose of clinical trial:

To compare hybrid closed-loop applying faster insulin aspart to hybrid closed-loop applying standard insulin aspart over 8 weeks.

Study objectives:

The study objective is to compare hybrid closed-loop glucose control using faster insulin aspart with hybrid closed-loop control using standard insulin aspart in very young children with type 1 diabetes.

1. EFFICACY: The objective is to assess the ability of a hybrid closed-loop system applying faster insulin aspart to maintain CGM glucose levels within the target range from 3.9 to 10.0 mmol/l, in comparison to a hybrid closed-loop system applying standard insulin aspart in very young children with type 1 diabetes.
2. SAFETY: The objective is to evaluate the safety of closed-loop glucose control using faster insulin aspart compared to standard insulin aspart in terms of episodes and severity of hypoglycaemia, frequency of diabetic ketoacidosis (DKA) and nature and severity of other adverse events.
3. UTILITY: The objective is to determine the acceptability and duration of use of the closed-loop system.
4. HUMAN FACTORS: The objective is to assess emotional and behavioural characteristics of parents/guardians and their response to the closed-loop system and clinical trial using validated surveys.

Participating clinical centres:

1. Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
2. John Radcliffe Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford
3. Nottingham Children's Hospital, Nottingham
4. Alder Hey Children's Hospital, Liverpool

Sample Size:

24 children randomised (6-14 participants per centre).

Maximum duration of study for a subject:

6 months

Recruitment:

Participants will be recruited through the paediatric diabetes outpatient clinics at participating clinical centres (see above). Enrolment will target up to 30 participants (aiming for 6-14 participants per centre), to allow for dropouts during run-in.

Consent:

Written informed consent will be obtained from all parents/guardians.

Screening and baseline Assessment:

Eligible participants will undergo a baseline assessment including a blood sample for the measurement of HbA1c. Height and weight will be recorded. Validated questionnaires will be completed by parents/guardians.

Pre-Study Training and Run-in:

Training sessions on the use of the study CGM, insulin pump and hybrid closed-loop insulin delivery will be provided by the research team. During the closed-loop training session, parents/guardians will operate the system under the supervision of the clinical research team. Participants and parents/guardians will use the study CGM, insulin pump, and hybrid closed-loop insulin delivery during a 2-4 week run-in period. For compliance and to assess the ability of the participant to use the study devices safely, at least 8 days of CGM data need to be recorded and safe use of study insulin pump and hybrid closed-loop insulin delivery demonstrated during the last 14 days of the run-in period. The CGM data will also be used to assess baseline glucose control and may be used for treatment optimisation as necessary.

Competency Assessment:

Competency on the use of study pump,study CGM and hybrid closed-loop insulin delivery will be evaluated by the research team. Training may be repeated if required.

Randomisation:

Eligible participants will be randomised using randomisation software to the initial use of faster insulin aspart with the hybrid closed-loop system or to standard insulin aspart with the hybrid closed-loop system for 8 weeks before crossing over to the other treatment arm.

1. Faster insulin aspart with hybrid closed-loop:

   Participants and their parents/guardians will use the hybrid closed-loop system with faster insulin aspart for 8 weeks at home. The participant, parents/guardians and the research team will be blinded to the intervention.

   Crossover assessment:

   At the end of the first study arm, validated questionnaires will be completed by the parents/guardians.
2. Standard insulin aspart with hybrid closed-loop:

Participants and their parents/guardians will use the hybrid closed-loop system with standard insulin aspart for 8 weeks at home. The participant, parents/guardians and the research team will be blinded to the intervention.

Study contacts:

Participants and parents/guardians will be contacted 24 hours after starting each study arm to ensure there are no concerns regarding the study devices. Participants will be contacted by the study team (email/phone) 2 and 4 weeks after the start of each study arm in order to record any adverse events, device deficiencies, and changes in insulin settings, other medical conditions and/or medication.

In case of any problems related to the technical devices or diabetes management, participants and parents/guardians will be able to contact a 24-hour telephone helpline to the local research team. The local research team will have access to central 24 hour advice on technical issues.

End of study assessments:

Height and weight will be recorded. Validated questionnaires will be completed by parents/guardians. Participants will resume usual care using their pre-study insulin pump.

Procedures for safety monitoring during trial:

Standard operating procedures for monitoring and reporting of all adverse events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.

A data safety and monitoring board (DSMB) will be informed of all serious adverse events and any unanticipated serious adverse device effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of subjects on safety grounds:

A participant and parent/guardian may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a participant after consideration of the benefit/risk ratio. Possible reasons are:

1. Serious adverse events
2. Serious protocol violation
3. Non-compliance
4. Failure to satisfy competency assessment
5. Decision by the investigator, or the Sponsor, that termination is in the participant's best medical interest
6. Allergic reaction to insulin

ELIGIBILITY:
Inclusion Criteria:

1. Age between 2 and 6 years (inclusive)
2. Type 1 diabetes as defined by WHO for at least 6 months [WHO definition: 'The aetiological type named type 1 encompasses the majority of cases which are primarily due to beta-cell destruction, and are prone to ketoacidosis. Type 1 includes those cases attributable to an autoimmune process, as well as those with beta-cell destruction for which neither an aetiology nor a pathogenesis is known (idiopathic). It does not include those forms of beta-cell destruction or failure to which specific causes can be assigned (e.g. cystic fibrosis, mitochondrial defects, etc.).']
3. Insulin pump user (with or without continuous glucose monitoring or flash glucose monitoring system) for at least 3 months, with parent/guardian good knowledge of insulin self-adjustment as judged by the investigator
4. Treated with U-100 rapid or ultra-rapid acting insulin analogue
5. Screening HbA1c ≤ 11% (97mmol/mol) on analysis from local laboratory
6. Able to wear glucose sensor
7. Able to wear closed-loop system 24/7
8. The parent/guardian is willing to follow study specific instructions
9. The parent/guardian is proficient in English

Exclusion Criteria:

1. Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
2. Untreated coeliac disease or thyroid disease based on local investigations prior to study enrolment
3. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids
4. Known or suspected allergy to insulin
5. Parent/guardian's lack of reliable telephone facility for contact
6. Parent/guardian's severe visual impairment
7. Parent/guardian's severe hearing impairment
8. Medically documented allergy towards the adhesive (glue) of plasters or subject is unable to tolerate tape adhesive in the area of sensor placement
9. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located in parts of the body which could potentially be used for localisation of the glucose sensor)

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Time in target (3.9 to 10.0mmol/L) (70 to 180 mg/dL) | 8-week intervention
  Time spent in the target glucose range from 3.9 to 10.0 mmol/l based on subcutaneous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Time spent above target glucose (10.0 mmol/L) (180 mg/dL) | 8-week intervention
  Percentage of time spent with sensor glucose readings above target glucose (10.0mmol/L) (180mg/dL)
Mean glucose | 8-week intervention
  Average of sensor glucose levels
Time spent below target glucose (3.9 mmol/L) (70 mg/dL) | 8-week intervention
  Percentage of time spent with sensor glucose readings below target glucose (3.9mmol/L)(70mg/dL)
Standard deviation of glucose | 8-week intervention
  Standard deviation Standard deviation of sensor glucose levels
Coefficient of variation of glucose | 8-week intervention
  Coefficient of variation of sensor glucose levels
Time spent below target glucose (3.0 mmol/L) (54 mg/dL) | 8-week intervention
  Percentage of time spent with sensor glucose readings below target glucose (3.0mmol/L)(54mg/dL)
Time with glucose levels in significant hyperglycaemia (glucose levels > 16.7 mmol/L) (300 mg/dL) | 8-week intervention
  Percentage of time spent with glucose levels in significant hyperglycaemia (glucose levels > 16.7mmol/L) (300mg/dL)
BMI SDS | 8-week intervention
Total, basal, and bolus insulin dose | 8-week intervention
Number of episodes of severe hypoglycaemia | Through study completion, an average of 5 months
  Safety evaluation
Frequency of diabetic ketoacidosis | Through study completion, an average of 5 months
  Safety evaluation
Frequency and nature of other adverse events or serious adverse events | Through study completion, an average of 5 months
  Safety evaluation
Closed-loop use | Through study completion, an average of 5 months
  Percentage of time of closed-loop is operational (Utility evaluation)
CGM use | Through study completion, an average of 5 months
  Percentage of time CGM is available (Utility evaluation)
Human factors assessment | 8-week intervention and 8-week control period
  Assessment of emotional and behavioural characteristics of parents/guardians, their response to the closed-loop system and information about parent/guardian sleep will be assessed through validated surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Study Director — Wellcome Trust-MRC Institute of Metabolic Science University of Cambridge
Locations (2):
- United Kingdom (2):
  - University Department of Paediatrics, Cambridge, Cambridgeshire
  - Wellcome Trust-MRC Institute of Metabolic Science University of Cambridge, Cambridge, Cambridgeshire

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.

REFERENCES:
- [Background] Tauschmann M, Thabit H, Bally L, Allen JM, Hartnell S, Wilinska ME, Ruan Y, Sibayan J, Kollman C, Cheng P, Beck RW, Acerini CL, Evans ML, Dunger DB, Elleri D, Campbell F, Bergenstal RM, Criego A, Shah VN, Leelarathna L, Hovorka R; APCam11 Consortium. Closed-loop insulin delivery in suboptimally controlled type 1 diabetes: a multicentre, 12-week randomised trial. Lancet. 2018 Oct 13;392(10155):1321-1329. doi: 10.1016/S0140-6736(18)31947-0. Epub 2018 Oct 3. PMID 30292578
- [Background] Tauschmann M, Allen JM, Nagl K, Fritsch M, Yong J, Metcalfe E, Schaeffer D, Fichelle M, Schierloh U, Thiele AG, Abt D, Kojzar H, Mader JK, Slegtenhorst S, Barber N, Wilinska ME, Boughton C, Musolino G, Sibayan J, Cohen N, Kollman C, Hofer SE, Frohlich-Reiterer E, Kapellen TM, Acerini CL, de Beaufort C, Campbell F, Rami-Merhar B, Hovorka R; KidsAP Consortium. Home Use of Day-and-Night Hybrid Closed-Loop Insulin Delivery in Very Young Children: A Multicenter, 3-Week, Randomized Trial. Diabetes Care. 2019 Apr;42(4):594-600. doi: 10.2337/dc18-1881. Epub 2019 Jan 28. PMID 30692242
- [Background] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Acerini CL, Dunger DB, Hovorka R. Home Use of Day-and-Night Hybrid Closed-Loop Insulin Delivery in Suboptimally Controlled Adolescents With Type 1 Diabetes: A 3-Week, Free-Living, Randomized Crossover Trial. Diabetes Care. 2016 Nov;39(11):2019-2025. doi: 10.2337/dc16-1094. Epub 2016 Sep 9. PMID 27612500
- [Background] Dovc K, Boughton C, Tauschmann M, Thabit H, Bally L, Allen JM, Acerini CL, Arnolds S, de Beaufort C, Bergenstal RM, Campbell F, Criego A, Dunger DB, Elleri D, Evans ML, Frohlich-Reiterer E, Hofer S, Kapellen T, Leelarathna L, Pieber TR, Rami-Merhar B, Shah VN, Sibayan J, Wilinska ME, Hovorka R; APCam11, AP@Home, and KidsAP Consortia. Young Children Have Higher Variability of Insulin Requirements: Observations During Hybrid Closed-Loop Insulin Delivery. Diabetes Care. 2019 Jul;42(7):1344-1347. doi: 10.2337/dc18-2625. Epub 2019 May 21. PMID 31221700
- [Background] Musolino G, Dovc K, Boughton CK, Tauschmann M, Allen JM, Nagl K, Fritsch M, Yong J, Metcalfe E, Schaeffer D, Fichelle M, Schierloh U, Thiele AG, Abt D, Kojzar H, Mader JK, Slegtenhorst S, Ashcroft N, Wilinska ME, Sibayan J, Cohen N, Kollman C, Hofer SE, Frohlich-Reiterer E, Kapellen TM, Acerini CL, de Beaufort C, Campbell F, Rami-Merhar B, Hovorka R; Kidsap Consortium. Reduced burden of diabetes and improved quality of life: Experiences from unrestricted day-and-night hybrid closed-loop use in very young children with type 1 diabetes. Pediatr Diabetes. 2019 Sep;20(6):794-799. doi: 10.1111/pedi.12872. Epub 2019 Jun 13. PMID 31140654
- [Derived] Ware J, Allen JM, Boughton CK, Cezar A, Hartnell S, Wilinska ME, Thankamony A, Deakin M, Leyland H, Phelan K, Thornborough K, Hovorka R. Hybrid Closed-Loop with Faster Insulin Aspart Compared with Standard Insulin Aspart in Very Young Children with Type 1 Diabetes: A Double-Blind, Multicenter, Randomized, Crossover Study. Diabetes Technol Ther. 2023 Jun;25(6):431-436. doi: 10.1089/dia.2023.0042. PMID 36880866